CLINICAL TRIAL: NCT02275195
Title: Immune Cell Dysfunction in Severe Alcoholic Hepatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B663
Record Dates: First submitted 2014-10-17; First posted 2014-10-27 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Hepatitis
Keywords: hepatitis; alcohol
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Through bio-sampling this study investigates the relationship between the frequency and function of the cells of a patients immune system and how these change and impact on the outcome of alcoholic hepatitis. the investigators will examine the role of different cells of the immune system and how they may determine the outcome of this condition. The investigators will also look at how established treatment strategies impact on the frequency and function of these cell subsets.

DETAILED DESCRIPTION:
Through bio-sampling this study investigates the relationship between the frequency and function of the cells of a patients immune system and how these change and impact on the outcome of alcoholic hepatitis. The investigators will examine the role of different cells of the immune system and how they may determine the outcome of this condition. The investigators will also look at how established treatment strategies impact on the frequency and function of these cell subsets.

Alcohol is the most common cause of liver disease in the developed world and results in the death of 2.5 million people annually. It is a causal factor in more than 60 major types of diseases and injuries and approximately 4.5% of the global burden of disease and injury is attributable to alcohol. Acute alcoholic hepatitis (AAH) is perhaps the most florid form of ALD and the leading cause of mortality in these patients is the development of sepsis which occurs in up to 40% of these patients and has a mortality rate of 50%.

By gaining a better understanding of the relationship between elements of the immune system and the progression to severe alcoholic hepatitis, it will allow the formulation of more effective treatment strategies for this condition.

Patients who agree to participate in this study will have an extra 40mls of blood drawn for scientific studies at the same time as routine blood samples are taken as part of their ongoing care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Patients presented with severe alcoholic hepatitis with a Maddrey score (discriminant function) of >32 (The Maddrey score uses various blood results on a patient to define the severity of alcoholic hepatitis e.g.bilirubin etc).
3. Ongoing abuse of alcohol (drinking in excess of 28 units/wk)

Exclusion Criteria:

1. Co-infection with HIV/Hepatitis B / Hepatitis C virus infection.
2. Patients with autoimmune liver disease.
3. Patients with metabolic liver disease.
4. Patients with significant psychiatric and/or neurological co-morbidity.
5. Hepatocellular carcinoma or other neoplastic disease
6. Pregnancy or breast feeding of infants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending / being treated at the Basildon Hospital for acute severe alcoholic hepatitis will be identified as potential participants in these studies
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To determine and changes to immune cell responses for outpatients with Alcoholic Hepatitis | Participants will be followed-up during thier hospital stay, which averages 4 weeks
  Characterize the relationship between various elements of patients immune system and the progression of an episode of severe Alcoholic Hepatitis

SECONDARY OUTCOMES:
Change from baseline to end of study in flow cytometry for patients with Alcoholic Hepatitis | on average 4 weeks
  Characterize the relationship between various elements of patients immune system and the progression of an episode of severe Alcoholic Hepatitis
Change from baseline to end of study in real time PCR for patients with Alcoholic Hepatitis | On average 4 weks
  Characterize the relationship between various elements of patients immune system and the progression of an episode of severe Alcoholic Hepatitis
Change from baseline to end of study in cell cultures for patients with Alcoholic Hepatitis | on average 4 weeks
  Characterize the relationship between various elements of patients immune system and the progression of an episode of severe Alcoholic Hepatitis

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Wright, MBBS MRCP, Principal Investigator — Basildon and Thurrock University Hospitals NHS FT
Locations (1):
- Basildon Hospital, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No